CLINICAL TRIAL: NCT00999505
Title: A Double-blind, Randomized, Placebo-controlled Trial With Amantadine as Adjunctive Therapy to Antipsychotics in Schizophrenia
Brief Title: Amantadine as Adjunctive Therapy to Antipsychotics in Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Clarissa Severino Gama, MD, PhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-303; 09-303
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Amantadine; Residual symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amantadine (Active Comparator): Amantadine 200mg twice a day
  Interventions: Drug: Amantadine
- Placebo (Placebo Comparator): Placebo capsules twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine — Amantadine 200mg twice a day over 12 weeks
  Other Names: Mantidan TM
  Arms: Amantadine
Drug: Placebo — Placebo capsules twice a day over 12 weeks
  Arms: Placebo

SUMMARY:
Amantadine as add-on therapy to antipsychotics may improve schizophrenia positive, negative and cognitive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Under antipsychotics with residual symptoms

Exclusion Criteria:

* Pregnancy
* Lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Scores in Brief Psychiatric Rating Scale | Baseline, 4 weeks, 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa S Gama, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil